CLINICAL TRIAL: NCT03660449
Title: A Prospective, Phase Ⅱ Study of S-1 Plus Moderately Hypofractionated Conformal Radiation for Esophageal Squamous Cell Carcinoma
Brief Title: Moderately Hypofractionated Conformal Radiation Combined With S-1 for Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1045
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Hypofractionated Conformal Radiation; S-1
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment (Experimental): All patients will receive two cycles of S-1 (40mg/㎡, BID, po) on D1-14, D22-35, combined with thoracic radiotherapy of 60 Gy/24 fractions for GTV and 40 Gy/16 fractions for CTV.
  Interventions: Combination Product: Moderately hypofractionated conformal radiation combined With S-1

INTERVENTIONS:
Combination Product: Moderately hypofractionated conformal radiation combined With S-1 — All patients will receive two cycles of S-1 (40mg/㎡, BID, po) on D1-14, D22-35, combined with thoracic radiotherapy of 60 Gy/24 fractions for GTV and 40 Gy/16 fractions for CTV.

SUMMARY:
This Phase II randomized study is to determine the efficacy and toxicities of moderately hypofractionated conformal radiation combined With S-1 for esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This Phase II randomized study is to determine the efficacy and toxicities of moderately hypofractionated conformal radiation combined With S-1 for esophageal squamous cell carcinoma.

All patients will receive two cycles of S-1 (40mg/㎡, BID, po) on D1-14, D22-35, combined with thoracic radiotherapy of 60 Gy/24 fractions for GTV and 40 Gy/16 fractions for CTV. The primary end point is progression-free survival, which is the time that passes from the first day of radiotherapy to the date on which disease progresses. Progression-free survival will be calculated and compared using the Kaplan-Meier method.Toxicities will be graded according to CTCAE v. 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal squamous cell carcinoma
* Inoperable stage II-IVa (UICC 2002; sixth edition), confirmed by contrast enhanced computed tomography,endoscopic ultrasonography, barium esophagram, emission computed tomography and/or positron emission tomography/computed tomography.
* Eastern Cooperative Oncology Group (ECOG) performance status 1-2
* Estimated life expectancy of at least 12 weeks
* Charlson comorbidity index.4
* Adequate bone marrow function: white blood cells grade 0 or 1,absolute neutrophils grade 0 or 1, platelets grade 0, haemoglobin grade 0 or 1
* Adequate renal function: creatinine grade 0 or 1
* Adequate liver function: serum bilirubin grade 0 or 1, alanine aminotransferase and aspartate aminotransferase <2 times of the upper normal limit
* Weight loss.15% during 6 months prior to diagnosis
* Forced expiratory volume second.1L

Exclusion Criteria:

* Prior history of malignancy, except for nonmelanoma skin carcinoma or cervical carcinoma in situ
* Previous anti-tumor therapy, including surgery, chemotherapy or radiotherapy
* Contraindication for chemotherapy or radiotherapy
* Malignant pleural or pericardial effusion
* Women in pregnancy or lactation period
* Women who has the probability of pregnancy without contraception
* Weight loss≥15% during 3 months prior to diagnosis
* In other clinical trials within 30 days
* Addicted in drugs or alcohol, AIDS patients
* Uncontrollable seizure or psychotic patients without self-control ability
* Severe allergy or idiosyncrasy
* Not suitable for this study judged by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 3 years

SECONDARY OUTCOMES:
Overall Survival | 3 years
rate of grade 3-4 radiation esophagitis | 1 year
rate of grade 3-4 radiation pneumonitis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Hui Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Background] Minsky BD, Pajak TF, Ginsberg RJ, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Kelsen DP. INT 0123 (Radiation Therapy Oncology Group 94-05) phase III trial of combined-modality therapy for esophageal cancer: high-dose versus standard-dose radiation therapy. J Clin Oncol. 2002 Mar 1;20(5):1167-74. doi: 10.1200/JCO.2002.20.5.1167. PMID 11870157
- [Background] Gaspar LE, Winter K, Kocha WI, Coia LR, Herskovic A, Graham M. A phase I/II study of external beam radiation, brachytherapy, and concurrent chemotherapy for patients with localized carcinoma of the esophagus (Radiation Therapy Oncology Group Study 9207): final report. Cancer. 2000 Mar 1;88(5):988-95. PMID 10699886
- [Background] Fan TY, Xing J, Lu J, Liu TH, Xu M, Zhang YJ, Shao Q, Li JB, Yu JM. Phase I/II study of induction chemotherapy plus concurrent chemotherapy and SMART-IMRT-based radiotherapy in locoregionally-advanced nasopharyngeal cancer. Oncol Lett. 2013 Mar;5(3):889-895. doi: 10.3892/ol.2013.1137. Epub 2013 Jan 15. PMID 23426016
- [Background] Koom WS, Kim TH, Shin KH, Pyo HR, Kim JY, Kim DY, Yoon M, Park SY, Lee DH, Ryu JS, Jung YS, Lee SH, Cho KH. SMART (simultaneous modulated accelerated radiotherapy) for locally advanced nasopharyngeal carcinomas. Head Neck. 2008 Feb;30(2):159-69. doi: 10.1002/hed.20667. PMID 17764088
- [Background] Butler EB, Teh BS, Grant WH 3rd, Uhl BM, Kuppersmith RB, Chiu JK, Donovan DT, Woo SY. Smart (simultaneous modulated accelerated radiation therapy) boost: a new accelerated fractionation schedule for the treatment of head and neck cancer with intensity modulated radiotherapy. Int J Radiat Oncol Biol Phys. 1999 Aug 1;45(1):21-32. doi: 10.1016/s0360-3016(99)00101-7. PMID 10477002
- [Background] Welsh J, Palmer MB, Ajani JA, Liao Z, Swisher SG, Hofstetter WL, Allen PK, Settle SH, Gomez D, Likhacheva A, Cox JD, Komaki R. Esophageal cancer dose escalation using a simultaneous integrated boost technique. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):468-74. doi: 10.1016/j.ijrobp.2010.10.023. Epub 2010 Dec 1. PMID 21123005
- [Background] Porceddu SV, Rosser B, Burmeister BH, Jones M, Hickey B, Baumann K, Gogna K, Pullar A, Poulsen M, Holt T. Hypofractionated radiotherapy for the palliation of advanced head and neck cancer in patients unsuitable for curative treatment--"Hypo Trial". Radiother Oncol. 2007 Dec;85(3):456-62. doi: 10.1016/j.radonc.2007.10.020. Epub 2007 Nov 26. PMID 18036689
- [Background] Agarwal JP, Nemade B, Murthy V, Ghosh-Laskar S, Budrukkar A, Gupta T, D'Cruz A, Pai P, Chaturvedi P, Dinshaw K. Hypofractionated, palliative radiotherapy for advanced head and neck cancer. Radiother Oncol. 2008 Oct;89(1):51-6. doi: 10.1016/j.radonc.2008.06.007. Epub 2008 Jul 21. PMID 18649963
- [Background] Hama Y, Uematsu M, Shioda A, Suda A, Aida S, Kusano S. Severe complications after hypofractionated high dose rate intracavitary brachytherapy following external beam irradiation for oesophageal carcinoma. Br J Radiol. 2002 Mar;75(891):238-42. doi: 10.1259/bjr.75.891.750238. PMID 11932217
- [Background] Aggarwal A, Harrison M, Glynne-Jones R, Sinha-ray R, Cooper D, Hoskin PJ. Combination external beam radiotherapy and intraluminal brachytherapy for non-radical treatment of oesophageal carcinoma in patients not suitable for surgery or chemoradiation. Clin Oncol (R Coll Radiol). 2015 Jan;27(1):56-64. doi: 10.1016/j.clon.2014.09.001. Epub 2014 Oct 11. PMID 25306490
- [Background] Song YP, Ma JB, Hu LK, Zhou W, Chen EC, Zhang W. Phase I/II study of hypofractioned radiation with three-dimensional conformal radiotherapy for clinical T3-4N0-1M0 stage esophageal carcinoma. Technol Cancer Res Treat. 2011 Feb;10(1):25-30. doi: 10.7785/tcrt.2012.500176. PMID 21214285
- [Background] Ma JB, Wei L, Chen EC, Qin G, Song YP, Chen XM, Hao CG. Moderately hypofractionated conformal radiation treatment of thoracic esophageal carcinoma. Asian Pac J Cancer Prev. 2012;13(8):4163-7. doi: 10.7314/apjcp.2012.13.8.4163. PMID 23098423
- [Background] Sato Y, Takayama T, Sagawa T, Okamoto T, Miyanishi K, Sato T, Araki H, Iyama S, Abe S, Murase K, Takimoto R, Nagakura H, Hareyama M, Kato J, Niitsu Y. A phase I/II study of nedaplatin and 5-fluorouracil with concurrent radiotherapy in patients with esophageal cancer. Cancer Chemother Pharmacol. 2006 Nov;58(5):570-6. doi: 10.1007/s00280-006-0193-x. Epub 2006 Feb 4. PMID 16463059
- [Background] Kodaira T, Fuwa N, Kamata M, Furutani K, Tachibana H, Yamazaki T. Single-institute phase I/II trial of alternating chemoradiotherapy with 5-FU and nedaplatin for esophageal carcinoma. Anticancer Res. 2006 Jan-Feb;26(1B):471-8. PMID 16739307
- [Background] Nemoto K, Matsushita H, Ogawa Y, Takeda K, Takahashi C, Britton KR, Takai Y, Miyazaki S, Miyata T, Yamada S. Radiation therapy combined with cis-diammine-glycolatoplatinum (Nedaplatin) and 5-fluorouracil for untreated and recurrent esophageal cancer. Am J Clin Oncol. 2003 Feb;26(1):46-9. doi: 10.1097/00000421-200302000-00010. PMID 12576924
- [Background] Tepper J, Krasna MJ, Niedzwiecki D, Hollis D, Reed CE, Goldberg R, Kiel K, Willett C, Sugarbaker D, Mayer R. Phase III trial of trimodality therapy with cisplatin, fluorouracil, radiotherapy, and surgery compared with surgery alone for esophageal cancer: CALGB 9781. J Clin Oncol. 2008 Mar 1;26(7):1086-92. doi: 10.1200/JCO.2007.12.9593. PMID 18309943
- [Derived] Zhou R, Luo G, Guo S, Wu Y, Luo Q, Wang D, Chen N, Liu F, Guo J, Ye W, Qiu B, Liu H. Moderately hypo-fractionated radiotherapy combined with S-1 in inoperable locally advanced esophageal squamous cell carcinoma: A prospective, single-arm phase II study (GASTO-1045). Front Oncol. 2023 Mar 10;13:1138304. doi: 10.3389/fonc.2023.1138304. eCollection 2023. PMID 36969023